CLINICAL TRIAL: NCT03150953
Title: Evaluation of a Novel Patient Warming System During MRI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Andrew Matisoff (Other)
Responsible Party: Sponsor-Investigator, Andrew Matisoff, MD, Children's National Research Institute
Organization: Children's National Research Institute (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 6559
Record Dates: First submitted 2017-05-10; First posted 2017-05-12 (Actual); Last update posted 2019-03-28 (Actual); Status verified 2019-03

CONDITIONS: Anesthesia; Hypothermia; Congenital Heart Disease
Keywords: anesthesia; MRI; thermoregulation
MeSH Terms: conditions — Hypothermia; Heart Defects, Congenital

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Standard of Care (No Intervention): Patients will receive standard of care which is 1-2 warm blankets.
- MRI-safe warming device (Experimental): The MRI-safe bore covering consists of a clear covering sheet positioned over the openings of the MRI scanner.
  Interventions: Device: MRI-safe bore covering
- MRI-safe warming device and Bair hugger (Experimental): IN addition to positioning the MRI-safe bore covering over the opening of the MRI scanner, the opening of the covering sheet will be connected to a device which blows warm air called a Bair Hugger. The Bair Hugger is an approved device, and MRI safe.
  Interventions: Device: MRI-safe bore covering

INTERVENTIONS:
Device: MRI-safe bore covering
  Arms: MRI-safe warming device; MRI-safe warming device and Bair hugger

SUMMARY:
Patients under deep sedation and general anesthesia lose heat to their surrounding environment. Hypothermia after anesthesia is associated with worse patient outcomes, including increased number of infections and cardiovascular complications. Cardiac MRI scans performed for patients who require general anesthesia can cause a loss of body heat.

Several mechanisms exist for reducing hypothermia under anesthesia including forced air warmers, fluid warmers, radiant warmers, and chemical warmers. Unfortunately, there are no MRI-compatible systems which allow patient warming and prevention of hypothermia in anesthetized patient in the MRI-scanner.

This study is testing a non-invasive device that warms patients under clinically indicated general anesthesia in the MRI scanner. This device will keep in the heat made by the MRI scanner.

DETAILED DESCRIPTION:
A. Each group will receive the usual clinical care for having an MRI under general anesthesia:

1. General anesthesia. The type of anesthesia used will be determined by the individual anesthesiologist, and will be the safest technique possible to allow for the desired MRI images to be obtained.
2. All participants will be covered with 1-2 warm blankets before receiving anesthesia and while in the scanner as part of standard warming measures.
3. All participants will have continuous temperature monitoring during the scan.

B. Participants will be randomized to one of the three

1. 20 subjects will receive the standard of care which is 1-2 warm blankets. This group is called the control group.
2. 20 study subjects will have the MRI-safe bore covering applied. This includes a clear covering sheet positioned over the openings of the MRI scanner.
3. 20 study subjects will have the MRI-safe bore covering applied, and in addition one opening of the covering sheet will be connected to a "Bair hugger" ( an approved device which blows warm air). The second opening will act as a vent to let air out of the MRI scanner bore. The Bair hugger will be programmed to deliver forced air at 38 degrees Celsius (approximately 100 degrees Fahrenheit) into the contained space within the MRI scanner.

Body temperature will be monitored continuously and documented in the electronic anesthesia record. The temperature of the forced air will be adjusted to maintain a goal body temperature of 36-38 degrees Celsius (96.8- 100.4 degrees Fahrenheit).

Image quality will be evaluated by the MRI-technologist and MRI -cardiologist subjectively.

ELIGIBILITY:
Inclusion Criteria:

1. Children < 7 years of age.
2. Undergoing medically necessary cardiovascular MRI under general anesthesia

Exclusion Criteria:

1.Patients with fever (temperature >38.5 degrees Celsius) or condition which require active cooling at the time of MRI

Max Age: 7 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Actual)
Dates: Start 2016-05-26 (Actual); Primary Completion 2018-05-01 (Actual); Study Completion 2018-11-30 (Actual)

PRIMARY OUTCOMES:
Normothermia maintenance using the MRI safe warming device | 15 minutes
  Body temperature will be monitored by either an esophageal stethoscope if patient is intubated or axillary temperature probe in patients who will undergo anesthesia without the need for an endotracheal tube. Temperature will be taken prior to being intubated or start of sedation, every 15 minutes, and at end of procedure when patient has returned to the recovery room.

SECONDARY OUTCOMES:
Quality of MRI images when using the MRI safe warming device | 90 minutes
  Images will be subjectively evaluated by the MRI technologist and MRI cardiologist for clarity.

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Matisoff, MD, Principal Investigator — Children's National Research Institute
Locations (1):
- Children's National Health System, Washington D.C., District of Columbia, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Diaz M, Becker DE. Thermoregulation: physiological and clinical considerations during sedation and general anesthesia. Anesth Prog. 2010 Spring;57(1):25-32; quiz 33-4. doi: 10.2344/0003-3006-57.1.25. PMID 20331336
- [Background] Reynolds L, Beckmann J, Kurz A. Perioperative complications of hypothermia. Best Pract Res Clin Anaesthesiol. 2008 Dec;22(4):645-57. doi: 10.1016/j.bpa.2008.07.005. PMID 19137808
- [Background] Manning W, Pennell D. Cardiovascular magnetic resonance. London: Churchill Livingstone; 2002.
- [Background] Balaban RS, Faranesh AZ, Hansen MS, Lederman RJ, Ratnayaka K. MRI scanner to infant incubator kit. Assignee: NIH. Provisional filed 2013. Tracking number: E-026-2013/0-US-01. Patent
- [Background] Kellman P, McVeigh ER. Image reconstruction in SNR units: a general method for SNR measurement. Magn Reson Med. 2005 Dec;54(6):1439-47. doi: 10.1002/mrm.20713. PMID 16261576